CLINICAL TRIAL: NCT00399971
Title: Phase I/II Study of An Ex Vivo Immunotherapy for Treatment of Idiopathic Aplastic Anemia
Brief Title: Safety and Efficacy Study of Ex Vivo Immunotherapy for Treatment of Aplastic Anemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Zhongxing Yangfan Biotech Co. Ltd. (Industry)
Collaborators: The 12th Guangzhou Municipal Hospital (Unknown); Liu Hua Qiao Hospital (Unknown)
Responsible Party: Demao Yang/Chief Scientist, Zhongxing Yangfan Biotech Co. Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAFocus
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Anemia, Aplastic
Keywords: Idiopathic Aplastic Anemia; Has Failed Conventional Immunosuppressive Therapy; Not Eligible For Bone Marrow Transplantation; C15.378.071.085
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hemathera (Experimental): Patients will receive cell-based immunotherapy.
  Interventions: Procedure: Ex Vivo Immunotherapy; Drug: Ex vivo immunotherapy

INTERVENTIONS:
Procedure: Ex Vivo Immunotherapy — Allogeneic and autologous ex vivo activated immune cells are given intravenously at least once a week
  Other Names: Aplastic Anemia, ex vivo Immunotherapy
Drug: Ex vivo immunotherapy — i.v. infusions, once a week, at least 6 to 12 months
  Other Names: Aplastic Anemia, ex vivo Immunotherapy

SUMMARY:
Our hypothesis is that ex vivo activated immune cells would produce multiple known and unknown potent hematopoietic cytokines, working in concert, these cytokines help stem cell growth and differentiation. Additionally, these cells travel and home to bone marrow as well as spleen and liver involved in hematopoietic activities, where direct cell-cell contact may be beneficial.

DETAILED DESCRIPTION:
Patients will be required to stay in our hospitals to receive the immunotherapy. Allogeneic peripheral blood mononuclear cells from healthy donors and the autologous peripheral mononuclear cells will alternately used for the treatment. Patients are expected to spend at least 6 to 12 months in the hospital and won't be released until they have improved significantly.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Idiopathic Aplastic Anemia
* Not Eligible for Bone Marrow Transplantation
* Not Responsive to Conventional Immunosuppressive Therapy

Exclusion Criteria:

* Leukemia or MDS or PNH or Fanconi's Disease
* pregnancy
* Allergic to Blood Product
* Severe Hypertension or Heart Disease
* Liver or Kidney Disease

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years

SECONDARY OUTCOMES:
Hematological Parameters | 2 years
Hematopoietic Activities in Bone Marrow | 2 years
Quality of Life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Demao Yang, PhD, Study Chair — Shenzhen Zhongxing Yangfan Biotech Co. Ltd.
Locations (1):
- Department of Hematology, Liu Hua Qiao Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen J, Liu W, Wang X, Chen H, Wu J, Yang Y, Wu L, Yang D. Ex vivo immunotherapy for patients with benzene-induced aplastic anemia. J Hematother Stem Cell Res. 2003 Oct;12(5):505-14. doi: 10.1089/152581603322448213. PMID 14594507
- [Background] Li G, Wang X, Wu L, Zhang W, Chen H, Xie Y, Yang D. Ex vivo activated immune cells promote survival and stimulate multilineage hematopoietic recovery in myelosuppressed mice. J Immunother. 2005 Jul-Aug;28(4):420-5. doi: 10.1097/01.cji.0000170360.99714.3f. PMID 16000962